CLINICAL TRIAL: NCT02090569
Title: ULtrasound Imaging in Focal Cortical dYSplasia: a New Approach to Delineating the Dysplastic Cortex During Neurosurgery
Brief Title: High Resolution Imaging of Cerebral Vasculature by Functional Micro-Doppler Sonography During Brain Surgery
Acronym: ULYS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: recommandation of the Data Safety monitoring Board
Sponsor: Centre Hospitalier St Anne (Other)
Collaborators: Fondation de l'Avenir (Other); Fondation pour les Sciences du Cerveau (Unknown); Association NEUROREFS (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D13-P007; 2013-A01231-44 (Other: ANSM)
Record Dates: First submitted 2014-01-28; First posted 2014-03-18 (Estimated); Last update posted 2018-01-25 (Actual); Status verified 2017-10

CONDITIONS: Partial Drug-resistant Epilepsy
Keywords: Functional micro-Doppler Sonography, fmDS, dysplasia, epilepsy, neurosurgery, cerebral blood volume, echography, hemodynamics
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Functional micro-Doppler sonography (Experimental)
  Interventions: Device: Functional micro-Doppler Sonography (fmDS)

INTERVENTIONS:
Device: Functional micro-Doppler Sonography (fmDS) — 1. Craniotomy according to MRI images
  2. Dura opening
  3. Sulcal Localization using neuronavigation
  4. Functional micro-Doppler Sonography including morphologic (Bmode) and functional measurement of the cerebral blood volume dynamics at high spatio-temporal resolution (100µm-20ms) using high-frequency (15MHz) ultrasound. At least 5 2-minute periods of spontaneous data will be recorded with a sampling rate for data acquisition of 15KHz and highpass filter of 10 to 70 Hz.
  5. Exeresis of the dysplasic tissue
  6. Control using fmDS before wound closure
  Other Names: DFC2 removal

SUMMARY:
High Resolution Imaging of Cerebral Vasculature by Functional Micro-Doppler Sonography During Brain Surgery (ULYS)

DETAILED DESCRIPTION:
Three decades since its comprehensive description (Taylor et al., 1971), focal cortical dysplasia (FCD) remains an enigmatic condition. FCD may cause severe refractory epilepsy that can be directly life threatening. Preoperative neuroimaging usually includes high-resolution MR imaging, which can reveal only 60 to 80% of cortical abnormalities in patients with FCD. When antiepileptic drugs fail to bring complete seizure freedom in FCD patients, surgical resection of the FCD is inevitable. Many patients, especially those with normal MR imaging results, undergo additional diagnostic procedures. Scalp EEG is frequently used and was one of the more important modalities during early surgical series. Approximately one half to two thirds of patients with abnormal EEG findings have a regional ictal abnormality. In some cases, intracranial electrophysiological recordings, most commonly with grid arrays, are used. Chronic recording allows identification of eloquent cortex areas, in addition to defining the epileptogenic region. The "eloquent brain" refers to the parts of the brain that allows the interaction with and the process of surrounding environment, via the senses, motion, language, memory and the purposeful use of tools. Nevertheless, all these techniques are either invasive or have a spatiotemporal resolution too poor to identify precisely the epileptic lesion deep in the brain. Hence, large resection of lesion areas, such as lobectomies and even hemispherectomies, are performed with a high risk of side effects including aphasia, partial face paralysis and hemiplegia depending on the localization of the lesion.

Navigable three-dimensional (3D)-MRI (based on Neuronavigation system) is currently used at the Sainte Anne hospital for planning and guiding during resection but neurosurgeons often complains about poor resolution and non-real-time imaging. While the use of surgical navigation has been an important advance in brain surgery, its utility is limited by the phenomenon known as brain shift. Whenever the brain is exposed, cerebral spinal fluid (CSF) is lost. Additionally, after the start of resectioning, the position of the surgical field can shift by centimeters, compared to the pre-surgery position. Brain shift makes it potentially hazardous to rely on preoperative images to determine the location of residual tumors. The only way to deal with brain shift and maintain accurate neuronavigation is with intraoperative imaging to enhance resection of the pathologic tissue in FCD.

Previously, the investigators demonstrated the feasibility of their approach by monitoring the hemodynamic responses during drug-induced epileptic seizures in preclinical models using functional micro-Doppler Sonography (fmDS).

The investigators are now developing this new tool combining a navigable three-dimensional (3D)-ultrasound interface to correct in real-time the brain shift (B-mode) with the near-real-time identification with unprecedented resolution of the dysplasia foci based on the specific hemodynamic signature of abnormal neurons.

ELIGIBILITY:
Inclusion Criteria:

* Age between 6 and 65 years
* Patient follow-up in the Neurosurgery department for a partial drug-resistant epilepsy
* Etiological diagnosis certain or likely of DCF2
* Operating indication
* consent (or agreement of the legal representative) to participate in the study

Exclusion Criteria:

* Etiological diagnosis other than a DCF2
* Refusal of consent
* No health insurance

Ages: 6 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2014-04-07 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Precise delineating of the dysplasic tissue in the white matter of patient with MRI-visible FCD using a 2D voxel-by-voxel analysis based on ultrasound B-Mode and micro-Doppler mode. | During the surgery at t0

SECONDARY OUTCOMES:
Determine if the location of abnormal dysplasic tissue correlate with location of the epileptogenic zone in MRI-visible FCD | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Bertrand DEVAUX, MD, PhD, Principal Investigator — Centre Hospitalier St Anne
Locations (1):
- Centre Hospitalier St Anne, Paris, France

REFERENCES:
- [Result] Mellerio C, Labeyrie MA, Chassoux F, Roca P, Alami O, Plat M, Naggara O, Devaux B, Meder JF, Oppenheim C. 3T MRI improves the detection of transmantle sign in type 2 focal cortical dysplasia. Epilepsia. 2014 Jan;55(1):117-22. doi: 10.1111/epi.12464. Epub 2013 Nov 15. PMID 24237393
- [Result] Mellerio C, Labeyrie MA, Chassoux F, Daumas-Duport C, Landre E, Turak B, Roux FX, Meder JF, Devaux B, Oppenheim C. Optimizing MR imaging detection of type 2 focal cortical dysplasia: best criteria for clinical practice. AJNR Am J Neuroradiol. 2012 Nov;33(10):1932-8. doi: 10.3174/ajnr.A3081. Epub 2012 May 3. PMID 22555587